CLINICAL TRIAL: NCT04315285
Title: Determining Optimal Verbal Instruction to Improve Walking Ability in People With Parkinson's Disease
Brief Title: Optimal Verbal Instruction to Improve Walking for PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201912096RIND
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Transcranial magnetic stimulation; Verbal instruction; Focus of attention; Parkinson's disease; Gait training
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher(s) who will conduct the outcome assessments will be masked from the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Active Comparator): 12 sessions of treadmill training with instruction of 'swing your arms'
  Interventions: Behavioral: Treadmill gait training with verbal instruction
- Heel-strike group (Experimental): 12 sessions of treadmill training with instruction of 'strike the ground with your heel'
  Interventions: Behavioral: Treadmill gait training with verbal instruction
- Big step group (Experimental): 12 sessions of treadmill training with instruction of 'lift your foot up high'
  Interventions: Behavioral: Treadmill gait training with verbal instruction
- Internal focus heel-strike (Experimental): 12 sessions of treadmill training with instruction of 'strike the ground with your heel'
  Interventions: Behavioral: Treadmill gait training with verbal instruction
- External focus shoe-strike (Experimental): 12 sessions of treadmill training with instruction of 'strike the ground with your shoe-heel'
  Interventions: Behavioral: Treadmill gait training with verbal instruction

INTERVENTIONS:
Behavioral: Treadmill gait training with verbal instruction — Each participant will receive 12 treatment with special verbal instruction which depends on participant's group. Each training session will last 60 minutes, including 5 minutes of warm-up stretching exercise, 40 minutes of treadmill training, and 15 minutes of over-ground gait and balance training. Throughout the 40 minutes of treadmill walking, the participants will walk on the level of 0% slope with a body-weight support system (LikorallTM 200, Liko, Sweden) used to protect the participants from falling; no actual weight support of the body will be provided. The frequency of intervention will be 2-3 days a week, spread across 4-6 weeks. The intervention protocols will be the same for all groups except the instruction provided to the participants in each group.

SUMMARY:
Background: One of the most disturbing motor symptoms in Parkinson's disease (PD) is gait disturbance. Clinicians often use various verbal instructions to correct abnormal gait patterns, and the most commonly used instruction is 'lift the foot up and make big steps.' Despite immediate performance improvement, people with PD are reluctant to walk outdoors with this exaggerated walking strategy because it makes them feel embarrassed, unbalanced, and fatigue easily. Since people with PD walk with flat foot, the investigators propose that an instruction emphasizing heel-strike at foot contact may be effective.

When delivering verbal instructions, clinicians should also consider the attentional focus of the instruction. Evidence has shown that instructions with external focus of attention (EF) is more beneficial than internal focus of attention (IF) for motor performance and learning. However, most of the gait-related instructions for PD are IF. The investigators thus aim to design a novel EF instruction and determine whether people with PD can benefit more from EF than IF instruction.

Objectives: (1) To investigate the effects of verbal instruction emphasizing heel-strike during gait training in people with PD. (2) To further determine whether an instruction with EF will induce greater training benefits than IF.

Methods: Two experiments will be conducted in this study. In experiment 1, 60 individuals with PD will be randomized into the heel-strike (HS), big-step (BIG), and control (CON) groups. All participants will receive 12 sessions of gait training with the specific verbal instruction allocated for each group. The participants will be assessed before, immediately after, and 4 weeks after the interventions. The primary outcome will be gait performance, and the secondary outcomes will include measurements of cognitive and behavioral functions. Additionally, transcranial magnetic stimulation will be used to examine the changes of corticomotor excitability associated with the interventions.

In the 2nd experiment, 46 individuals with PD will be randomized into the internal focus heel-strike (IF-HS) or external focus shoe-strike (EF-SS) group. Except for the verbal instruction provided to the participants, other intervention and testing procedures will be the same as experiment 1.

Group × time repeated measures analysis of variance (ANOVA) will be used to compare the intervention effects among the groups, and a significance level will be set at α=0.05.

DETAILED DESCRIPTION:
Background: One of the most disturbing motor symptoms in Parkinson's disease (PD) is gait disturbance. Clinicians often use various verbal instructions to correct abnormal gait patterns, and the most commonly used instruction is 'lift the foot up and make big steps.' Despite immediate performance improvement, people with PD are reluctant to walk outdoors with this exaggerated walking strategy because it makes them feel embarrassed, unbalanced, and fatigue easily. Since people with PD walk with flat foot, the investigators propose that an instruction emphasizing heel-strike at foot contact may be effective. The action of heel-strike could function as a foot rocker and facilitate forward progression of the limb. Heel-strike could also increase the effective limb length and reduce energy cost during walking. Thus, emphasizing heel-strike during gait training may restore near-normal gait pattern and enhance the patients' compliance.

When delivering verbal instructions, clinicians should also consider the attentional focus of the instruction. Evidence has shown that instructions with external focus of attention (EF) is more beneficial than internal focus of attention (IF) for motor performance and learning. However, most of the gait-related instructions for PD are IF. The investigators thus aim to design a novel EF instruction and determine whether people with PD can benefit more from EF than IF instruction.

Objectives: The first aim of this study is to investigate the effects of verbal instruction emphasizing heel-strike during gait training in people with PD. The second aim is to further determine whether an instruction with EF will induce greater training benefits than IF.

Methods: Two experiments will be conducted in this study. In experiment 1, 60 individuals with idiopathic PD will be randomized into the heel-strike (HS), big-step (BIG), and control (CON) groups. All participants will receive 12 sessions of treadmill and over-ground gait training. During training, the participants will be instructed to 'strike the ground with the heel,' 'lift the foot up high,' or 'swing the arms' in the HS, BIG, or CON group, respectively. The participants will be assessed before, immediately after, and 4 weeks after the interventions. The primary outcome will be gait performance, and the secondary outcomes will include finger sequence task, Montreal Cognitive Assessment test, Stroop Color-Word test, Unified Parkinson's Disease Rating Scale, 5 times sit to stand test, Timed Up and Go test, Fatigue Severity Scale, Activities-Specific Balance Confidence Scale, Parkinson's Disease Questionnaire-39, New Freezing of Gait Questionnaire and Geriatric Depression Scale. Transcranial magnetic stimulation will be used to examine the changes of corticomotor excitability associated with the interventions.

In the 2nd experiment, 46 individuals with PD will be randomized into the internal focus heel-strike (IF-HS) or external focus shoe-strike (EF-SS) group. The instruction for the IF-HS group will be 'strike the ground with the heel,' and 'strike the ground with the shoe-heel' for the EF-SS group. The other intervention and testing procedures will be the same as experiment 1.

Group × time repeated measures analysis of variance (ANOVA) will be used to compare the intervention effects. The partial eta square (η2) will be calculated to determine the magnitude of group differences. A significance level will be set at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* able to follow instructions to perform the tasks (Mini Mental State Examination ≥ 24)
* able to read and hear properly without or with aids (e.g., eyeglasses or hearing aids)
* can walk independently with or without devices

Exclusion Criteria:

* has other neurological disorders in addition to PD
* has deep brain stimulation or pacemaker implanted in their body
* has a family-history of epilepsy
* has a self-history of seizure
* has unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Gait performances | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The participants will be required to walk along a 5-meter walkway in their comfortable walking speed for 5 trials under single and dual-task walking conditions. The gait performances will be captured by the Physilog®5 system (Gait Up, Renens, Switzerland), which include two inertial sensors with built-in 3D accelerometers and gyroscopes.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The MoCA will be used to evaluate general cognitive function of the participants. It evaluates several cognitive functions including attention, set-shifting, short-term memory, verbal fluency, calculation, orientation, digit span, conceptual thinking, and visuospatial processing skills. The total score of MoCA is 30 with a higher score indicating better cognitive function. The MoCA has good to excellent psychometric properties
The Stroop Color-Word test | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The Stroop Color-Word test will be used to evaluate the changes in executive functions in people with PD. The executive functions involved in the Stroop Color-Word test are selective attention, inhibition, and set-shifting. The Stroop Color-Word test comprises the congruent and incongruent testing conditions. The congruent condition is when the color ink of a word is coherent with the written color name, and the incongruent condition is when the color ink differs from the written color name (e.g., the word 'red' written in blue ink). The participants are instructed to read out the ink color of the word, but not the color word name, as accurately and as fast as possible within 45 seconds.
The Unified Parkinson's Disease Rating Scale (UPDRS) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a well-established and widely used rating tool for the evaluation of disease severity of PD. The UPDRS consists of 4 sections: 1) Mentation, Behavior, and Mood, 2) Activities of daily living (ADL), 3) Motor examination, and 4) Complications of therapy. In this proposed study, we will only evaluate Part 3 of the scale - the motor disturbances of the patients. The section of "motor examination" contains 18 tests with 33 items (some tests contain movement of the left and right extremities and/or trunk), and each item scores from 0 (absent of the symptom) to 4 (marked in the symptom and present most of the time). The total score ranges from 0 to 132 for Part 3 of the UPDRS with a lower score indicates less PD symptoms and a higher score suggests more severe in PD disease. Internal consistency and validity has been established to be excellent for UPDRS.
Fatigue severity questionnaire (FSS) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The FSS will be used to determine how fatigue interferes an individual's daily living and social participation. It contains 9 items, and each item is scored on a 7-point scale with a score 1 indicates strongly disagree and score 7 indicates strongly agree. The total score ranges from 9 to 63, with a higher score indicate greater fatigue severity.
Parkinson's Disease Questionnaire-39 (PDQ-39) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The PDQ-39 is a self-report questionnaire containing 39 items assessing the impact of PD on quality of life. The PDQ-39 covers 8 dimensions: mobility, activities of daily living, emotional well-being, stigma, cognition, communication, and bodily discomfort. The participants are required to answer the questions based on their experiences in the preceding month prior to the interview. The scoring system for each item ranges from 0 (never have difficulty) to 4 (always have difficulty) with lower scores suggesting better quality of life.
New Freezing of Gait Questionnaire (NFOG-Q) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The NFOG-Q will be used to evaluate the freezing frequency and severity of the patients with PD. It composes of 3 parts; in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. PartⅡassesses the severity of FoG according to the frequency and duration of the freezing episodes, while PartⅢevaluates the impact of freezing on daily activities, such as walking. The reliability and internal consistency of the NFOG-Q have been well-established for patients with PD.
Geriatric Depression Scale (GDS) | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The GDS is a self-report measure of depression in older adults. The GDS contains 15 items, and the users respond in a "Yes/No" format to each question in reference to the past 1 week.
The Timed Up and Go (TUG) Test | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The participants will initially sit on a comfortable chair with hips and knees flexed at 90°. Upon a 'GO' signal, the participants will stand up from the chair, walk for 3 meters, turn around, walk back to the chair, and sit down. The participants will be instructed to complete the task at their preferred/ comfortable speed. Good to excellent test-retest reliability and inter-rater reliability have been established in people with PD.
Finger sequence task | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  A finger sequence task will be used to evaluate motor learning ability. The finger sequence task contains 3 numerical sequences, and each sequence is embedded with colored circles and presented on a specific location on the computer screen. The participants will not be informed about the specific sequence-context associations; they will only be instructed to use their index and middle finger of both hands to press the keys for the numerical sequences in a sequential order of 1-2-3-4 as accurately and as fast as possible. The 3 sequences will be presented on the computer screen in a pseudorandom order, and the participants will be required to complete a total of 324 trials (108 trials per sequence) during the acquisition period. Ten minutes and 24 hours after practice, the participants will be tested under different testing conditions.
Activities-Specific Balance Confidence (ABC) Scale | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The Activities-Specific Balance Confidence (ABC) scale will be used to examine an individual's confidence level of not falling when performing activities of daily living. The ABC Scale contains 16 different activities performed indoors and outdoors. The participants will be asked to rate their confidence level (range from 0% to 100% of confidence) of not falling for each item. An average score of the 16 items (range from 0% to 100%) will be calculated to determine the participant's confidence level of not falling when performing the activities of daily living. The internal consistency and test-retest reliability of the ABC scale in patients with PD were excellent.
Corticomotor excitability | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  Transcranial magnetic stimulation (TMS) will be used to evaluate corticomotor excitability. Corticomotor excitability outcomes will include resting motor threshold (RMT), motor evoke potential (MEP), cortical silent period (CSP) duration, short-interval intracortical inhibition (SICI), intracortical facilitation (ICF), and long-interval intracortical inhibition (LICI). The RMT could reflect the membrane excitability of the corticospinal neurons and the cortical interneurons. Peak-to-peak MEP amplitude is an indicator of the integrity and excitability of the corticospinal tract. The CSP is a period when EMG activity being suppressed for a few hundred milliseconds after the MEP, and has often been used as an indicator of the inhibitory mechanism occurs within the corticospinal tract. The SICI, ICF, and LICI have been identified to be good indicators of intracortical inhibition and facilitation.
Five Times Sit-to-Stand (FTSTS) Test | Three time points: pre-test(before intervention), post-test(immediate after intervention), follow-up test(one month after intervention)
  The FTSTS test will be evaluated to represent the strength and endurance of the lower limbs. The participants will be sat on a standardized chair, and they will be required to stand up and then sit down for 5 times as fast as possible. The amount of time the participants need to complete the task will be recorded, and a lesser amount of times would indicate better strength of the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Yun Lee, PhD, Principal Investigator — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, NTU, Taiwan, Taipei, Taiwan

REFERENCES:
- [Derived] Li MH, Tai CH, Luh JJ, Chen YJ, Hsu WL, Lee YY. Influence of Verbal Instruction on Gait Training in Parkinson Disease: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2024 Jul 1;103(7):617-623. doi: 10.1097/PHM.0000000000002420. Epub 2024 Jan 6. PMID 38207195